CLINICAL TRIAL: NCT06363344
Title: Study of the Implementation of a Post-hospitalization Follow-up Consultation in a Pediatric Intensive Care Unit: Needs, Acceptability, Cooperation
Brief Title: Follow-up in Pediatric Intensive Care Unit
Acronym: APRELAREA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP231022; IDRCB: 2023-A00660-45 (Registry Identifier: IDRCB ANSM)
Record Dates: First submitted 2024-01-31; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-01

CONDITIONS: Intensive Care Psychosis
Keywords: pediatrics; tertiary prevention; resuscitation; hospital organizational innovations; coordination
MeSH Terms: interventions — Patient Health Questionnaire

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multi professional and comprehensive management of patients (Other): An advanced practice nurse who is a member of the PICU team monitors patients. Contact with children and their family is established shortly before leaving intensive care, and the child and his family are seen again few days after by the nurse where the child was discharged, then closely in the 3 months following discharge (at 1 and 3 months).
  Interventions: Other: Questionnaires : PHQ-9 (Kroenke, 2001), the PSC (Sheldrick, 2012), the ASQ-SE (Squires, 2015), the PedsQL (Varni, 1999)

INTERVENTIONS:
Other: Questionnaires : PHQ-9 (Kroenke, 2001), the PSC (Sheldrick, 2012), the ASQ-SE (Squires, 2015), the PedsQL (Varni, 1999) — An advanced practice nurse who is a member of the PICU team monitors patients by questionnaires at 1 and 3 months. Depending on the anomalies detected, whether at the somatic, psychological, emotional or social level, the nurse refers to competent specialists and collaborators and continues monitoring of the family as needed.

SUMMARY:
Background In developed countries, mortality rates in pediatric intensive care units (PICUs) are around 4% and thus, most children admitted to these units survive. However, some pediatric survivors experience long-term morbidity (cognitive, psychological, social and/or physical disorders) associated with their intensive care stay. Currently in France, there are no recommendations for the management of these patients and most of them do not have standardized follow-up.

Objectives Main objective: To assess the feasibility of implementing systematic and comprehensive management of pediatric patients who have been admitted to the PICU.

Intermediate objectives are to study:

* The needs of the children and their families which should be met by this management
* The acceptability of this organizational innovation for all the actors involved
* The cooperation between actors of the hospital and city health system + social professionals involved
* The costs of implementation and the budgetary impact of such a system

Methods Needs assessment: questionnaires and interviews with patients and their families (parents and possibly siblings if involved) to collect the medico-psycho-social impact of the PICU stay at the time of discharge and 3 months later.

Study of acceptability: quantitative survey of health professionals involved in the care of these children and expected care modalities. This includes pediatric intensivists, professionals from the children's usual care services (if applicable), attending physician.

Study of cooperation: analysis of needs and of the network usually solicited for the children benefiting from this care: who is identified, who remains to be identified, obstacles. Quantitative analysis of consultation reports and survey of professionals.

Budgetary impact analysis: study of the cost of setting up consultations for the health care system, and study of its financial and health consequences for the main needs identified, on the basis of data from the literature and expert opinions

Perspectives Compare the benefit of this systematic, multi professional and comprehensive management of pediatric patients after PICU discharge versus standard of care

DETAILED DESCRIPTION:
Background In developed countries, mortality rates in pediatric intensive care units (PICUs) are around 4% and thus, most children admitted to these units survive. However, some pediatric survivors experience long-term morbidity (cognitive, psychological, social and/or physical disorders) associated with their intensive care stay. Currently in France, there are no recommendations for the management of these patients and most of them do not have standardized follow-up.

Objectives Main objective: To assess the feasibility of implementing systematic and comprehensive management of pediatric patients who have been admitted to the PICU.

Intermediate objectives are to study:

* The needs of the children and their families which should be met by this management
* The acceptability of this organizational innovation for all the actors involved
* The cooperation between actors of the hospital and city health system + social professionals involved
* The costs of implementation and the budgetary impact of such a system

Methods Needs assessment: questionnaires and interviews with patients and their families (parents and possibly siblings if involved) to collect the medico-psycho-social impact of the PICU stay at the time of discharge and 3 months later.

Study of acceptability: quantitative survey of health professionals involved in the care of these children and expected care modalities. This includes pediatric intensivists, professionals from the children's usual care services (if applicable), attending physician.

Study of cooperation: analysis of needs and of the network usually solicited for the children benefiting from this care: who is identified, who remains to be identified, obstacles. Quantitative analysis of consultation reports and survey of professionals.

Budgetary impact analysis: study of the cost of setting up consultations for the health care system, and study of its financial and health consequences for the main needs identified, on the basis of data from the literature and expert opinions

Perspectives Compare the benefit of this systematic, multi professional and comprehensive management of pediatric patients after PICU discharge versus standard of care

ELIGIBILITY:
Inclusion Criteria:

* All children discharged alive from the paediatric intensive care unit
* Hospitalized in paediatric intensive care unit for 3 days or more
* Parents and children agreeing to follow-up by the advanced practice nurse

Exclusion Criteria:

* Impromptu transfers (making it impossible to collect information the day before discharge) or death
* Intellectual retardation of child/parent preventing data collection by questionnaire
* Participant unable or unwilling to comply with study procedures (including those unable to speak French; those unable to honor a follow-up consultation within 3 months)

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Emotional and behavioral problem of the children measured by the PSC questionnaire (Sheldrick, 2012) | 24 months

SECONDARY OUTCOMES:
Mental disorders measured by the PHQ-9 (Kroenke, 2001) questionnaire | 24 months
Social-emotional development measured by the ASQ-SE (Squires, 2015) questionnaire | 24 months
Pediatric Quality of Life measured by the the PedsQL (Varni, 1999) questionnaire | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michaël LEVY, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided